CLINICAL TRIAL: NCT04505826
Title: A Phase I Dose Escalation and Dose Expansion and Phase II Monotherapy Open-label, First-in-Human, Multicenter Study of OP-1250 in Adult Subjects With Advanced and/or Metastatic Hormone Receptor (HR)-Positive, HER2-negative Breast Cancer
Brief Title: A Dose Escalation/Expansion Study of Oral OP-1250 in Subjects With Advanced and/or Metastatic HR+, HER2- Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Olema Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OP-1250-001
Record Dates: First submitted 2020-07-21; First posted 2020-08-10 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-07

CONDITIONS: Hormone Receptor Positive Breast Carcinoma; HER2-negative Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OP-1250 Phase I Part A (Dose Escalation) and Part B (Dose Expansion) (Experimental): Phase I Part A will evaluate the safety and pharmacokinetics (PK)of a range of OP-1250 doses to identify the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D). Phase I Part B will evaluate the safety and PK of OP-1250 to confirm the RP2D dose.
  Interventions: Drug: OP-1250
- OP-1250 Phase II (Experimental): This portion of the study further explores the clinical activity, safety, and PK of OP-1250 monotherapy at the RP2D and will estimate preliminary anti-tumor efficacy in 3 cohorts.
  Cohort A will enroll subjects with measurable disease without evidence of CNS metastases; Cohort B will enroll subjects with non-measurable (evaluable) disease without evidence of CNS metastases; and Cohort C will enroll subjects with evaluable disease (measurable and non-measurable) with CNS metastases.
  Interventions: Drug: OP-1250

INTERVENTIONS:
Drug: OP-1250 — Complete Estrogen Receptor ANtagonist (CERAN)

SUMMARY:
This clinical trial is a Phase I dose escalation and dose expansion and Phase II monotherapy open-label, first-in-human, multicenter study of OP-1250 in adult subjects with advanced and/or metastatic hormone receptor (HR)-positive, her2-negative breast cancer.

DETAILED DESCRIPTION:
This is a Phase I dose escalation and dose expansion and Phase II monotherapy open--label, first--in--human study to determine the dose limiting toxicity (DLT), maximum tolerated dose (MTD) and/or recommended Phase II dose (RP2D), to characterize the safety and pharmacokinetic (PK) profile, and to estimate the preliminary anti-tumor activity of OP-1250 as a single agent in adult subjects with hormone receptor (HR)-positive/human epidermal growth factor receptor 2 (HER2)-negative metastatic or locally advanced breast cancer. This study comprises 2 Phases: Phase I (Part A [Dose Escalation] and Part B [Dose Expansion]) and Phase II. Additionally, all subjects (Phase I and Phase II) will be eligible to participate in 1 of 2 sub-studies. Patients must have received at least 1 prior hormonal regimen and at least 6 months of a prior continuous endocrine therapy for locally advanced or metastatic disease. Patients will be evaluated for treatment emergent adverse events (AEs) during study participation, and toxicity will be assessed according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events, Version 5.0.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Must have received at least 1 prior hormonal regimen and at least 6 months of a prior continuous endocrine therapy for locally advanced or metastatic disease
* Must not have received prior oral endocrine therapy < 2 weeks prior to first dose
* Must not have received prior, chemotherapy in 2 weeks or within 5 half-lives whichever is earlier, antibody therapy within 4 weeks or investigational therapy within 4 weeks or 5 half-lives whichever is earlier, prior to the first dose
* Adequate hepatic function
* Adequate renal function
* Normal coagulation panel
* Willingness to use effective contraception

Exclusion Criteria:

* Gastrointestinal disease
* Significant renal disease
* Significant cardiovascular disease
* Significant ECG abnormalities
* Ongoing systemic bacterial, fungal, or viral infection (requiring antimicrobial therapy)
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | The first 28 days of treatment
  To determine the maximum tolerated dose (MTD) and/or recommended Phase II dose (RP2D) of OP-1250, the incidence of DLTs will be assessed.
Characterize the incidence, nature and severity of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) of OP-1250 | Up to 42 days after end of treatment
  Characterize the incidence, nature and severity of TEAEs and SAEs of OP-1250 according to NCI-CTCAE version 5.0
Pharmacokinetics of OP-1250 | Every 28 days
  Plasma concentrations of OP-1250 will be assessed at predefined intervals
Anti-tumor activity of OP-1250 | Every 8 weeks
  Tumor response will be evaluated in patients with measurable or evaluable disease, using RECISTv1.1 guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Mark Shilkrut, MD, Study Director — Olema Pharmaceuticals, Inc.
Locations (19):
- United States (15):
  - UCLA Hematology/Oncology, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - University of Miami, Sylvester Comprehensive Cancer Center, Deerfield Beach, Florida
  - Advent Health, Orlando, Florida
  - Florida Cancer Center, Sarasota, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Sarah Cannon Research Institute, Nashville, Tennessee
- Australia (4):
  - Macquarie University, Sydney, New South Wales
  - Westmead, Westmead, New South Wales
  - ICON Cancer Centre, Auchenflower, Queensland
  - Cancer Research South Australia, Adelaide, South Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hamilton EP, Patel MR, Borges VF, Meisel JL, Okera M, Alemany CA, Pluard TJ, Wesolowski R, Sabanathan D, Miller KD, Conlin AK, McCarthy N, Shaw M, Tonda M, Shilkrut M, Lin NU. Palazestrant, a novel oral Complete Estrogen Receptor Antagonist (CERAN) and Selective Estrogen Receptor Degrader (SERD), in patients with ER+/HER2- advanced or metastatic breast cancer: phase 1/2 study results. Breast Cancer Res. 2025 Jul 1;27(1):119. doi: 10.1186/s13058-025-02049-y. PMID 40598566